CLINICAL TRIAL: NCT02657616
Title: Stroke Prophylaxis of Patients With Atrial Fibrillation: Real-life Effectiveness and Safety of Novel Anticoagulants Compared to Vitamin-k-antagonists Based on an Analysis of German Claims Data
Brief Title: Stroke Prophylaxis of AF-patients: Real-life Effectiveness and Safety of Novel Anticoagulants Compared to VKA
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakoökonomie und Arzneimittellogistik e.V. (Other)
Responsible Party: Principal Investigator, Sabrina Müller, Principal investigator, Institut für Pharmakoökonomie und Arzneimittellogistik e.V.
Other Study IDs: NOAC001
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation; Stroke Prophylaxis
MeSH Terms: conditions — Atrial Fibrillation | interventions — acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- No anticoagulation with VKA/NOAC: No prescriptions of vitamin-k-antagonists/novel anticoagulants in all observational period; No prescriptions of low molecular weight heparins/Clopidogrel during observation period to the extent of more than 30 days.
- Anticoagulation with vitamin-k-antagonists: The patient should be treated stable during the observation period with vitamin-k-antagonists (at least one prescription per half-year). The patient should be not been around on other anticoagulants during the observation period. This means that no prescriptions of novel anticoagulants and not more than 30 days should be observable prescriptions of low molecular weight heparins/Clopidogrel per year.
  Interventions: Drug: vitamin-k-antagonists
- Anticoagulation with novel oral anticoagulants: The patient should be treated stable during the observation period with a novel anticoagulant (at least one prescription per half-year). This means that no vitamin-k-antagonists prescriptions and not more than 30 days should be observable prescriptions of low molecular weight heparins/Clopidogrel per year from the start of the observation period.
  Interventions: Drug: Novel oral anticoagulants

INTERVENTIONS:
Drug: vitamin-k-antagonists
  Groups: Anticoagulation with vitamin-k-antagonists
Drug: Novel oral anticoagulants
  Groups: Anticoagulation with novel oral anticoagulants

SUMMARY:
The central questions of the study can be summarized as follows:

What stroke / death rates are the result of the use of the following treatment strategies: no anticoagulation with vitamin-k-antagonists (VKAs) or novel oral anticoagulants (NOACs), anticoagulation with VKAs and anticoagulation with NOACs (all). What other thromboembolic complication rates resulting from the use of these treatment strategies? What heavy bleeding rates resulting from the defined management strategies? The analysis is based on a data set of patients with atrial fibrillation (AF)(01/01/2010 - 30/06/2014). 2010 is used as the reference period and 01/01/2011-30/06/2013 as the inclusion period. The minimum observation time per patient is 12 months.

Used is a data base of the AOK PLUS as well as the AOK Baden-Württemberg and AOK Bayern.

The aim of the study is to compare clinical outcomes between the different treatment strategies (frequency of events and time to first event). The influence of alternative treatment strategies is measured on the basis of three different methodological approaches: unadjusted comparison of event council and time to first event between the defined patient groups; matched-pair comparison (propensity score matching) between the different groups of patients (treatment strategies) and multivariate analysis using time to event (Cox proportional hazards model) as the dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* one inpatient or two outpatient confirmed diagnosis of atrial fibrillation in two different quarters
* Continuously insured by the AOK PLUS, AOK Bayern or AOK Baden-Württemberg

Exclusion Criteria:

* Age < 18 years
* Maximum possible observational period < 12 months (exception: death)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis is based on a data set of patients with atrial fibrillation (01/01/2010 - 30/06/2014) insured by the AOK PLUS, AOK Bayern or AOK Baden-Württemberg.
Sampling Method: Non-Probability Sample
Enrollment: 204464 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Death | 01/01/2011-30/06/2014; at least 12 months; up to 40 months
Transient ischemic attack | 01/01/2011-30/06/2014; at least 12 months; up to 40 months
Ischemic stroke | 01/01/2011-30/06/2014; at least 12 months; up to 40 months
Hemorrhagic stroke | 01/01/2011-30/06/2014; at least 12 months; up to 40 months
Heavy bleeding | 01/01/2011-30/06/2014; at least 12 months; up to 40 months

REFERENCES:
- [Derived] Mueller S, Groth A, Spitzer SG, Schramm A, Pfaff A, Maywald U. Real-world effectiveness and safety of oral anticoagulation strategies in atrial fibrillation: a cohort study based on a German claims dataset. Pragmat Obs Res. 2018 May 1;9:1-10. doi: 10.2147/POR.S156521. eCollection 2018. PMID 29750067